CLINICAL TRIAL: NCT05102565
Title: A Dyadic Telehealth Program to Support Alzheimer's Disease Patients and Their Caregivers During COVID-19
Brief Title: A Dyadic Telehealth Program for Alzheimer's Patients/Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Yeonsu Song, PhD, RN, FNP, Assistant Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K23AG055668-04S1 (NIH)
Record Dates: First submitted 2021-10-09; First posted 2021-11-01 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Sleep
Keywords: dementia; caregivers; COVID-19 pandemic
MeSH Terms: conditions — Dementia; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): 6 weekly sleep education program
  Interventions: Behavioral: sleep education program

INTERVENTIONS:
Behavioral: sleep education program — A multicomponent behavioral sleep program, consisting of sleep hygiene, stimulus control, sleep compression, pleasurable activity, daily walking, and light exposure.

SUMMARY:
This study aims to refine and evaluate feasibility of a telehealth intervention for persons with Alzheimer's disease and their caregivers. The intervention will use evidence-based techniques for decreasing symptoms of depression, anxiety, and poor sleep, that are commonly reported among this vulnerable group during the COVID-19 pandemic. Improved symptoms among this group may improve their other health outcomes and quality of life and furthermore the quality of care that caregivers provide for persons with Alzheimer's disease during this challenging time.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients

* Have a diagnosis of AD (probable or possible), other related dementia, or mild cognitive impairment as documented in electronic medical record
* Community-dwelling
* Aged > 50 years
* Have no previously diagnosed sleep disorders (e.g., sleep apnea, restless legs syndrome)
* Able to ambulate with or without assistive devices (i.e., dyads will be excluded if the care recipient is bedbound)
* Have an eligible caregiver

Inclusion criteria for caregivers

* Aged >18 years
* Live with the eligible patient
* Have regularly assisted the care recipient with >1 of 7 basic activities of daily living (ADLs; i.e., eating, dressing/undressing, grooming, walking across a room, getting in and out of bed, bathing, toileting) or >1 of 7 Instrumental ADL (IADLs; i.e., using the telephone, getting to places beyond walking distance, shopping, preparing meals, doing housework, taking medicine, handling money) for the past 6 months
* Have no history of cognitive impairment
* Can communicate in English.

Exclusion Criteria:

-Professional caregivers will be excluded. Patients will be excluded if they are bedbound. If the eligibility criteria for either a patient or a caregiver are not met, their dyads will be excluded for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Sleep efficiency-Actigraphy | immediately after the last session of the intervention
  Nighttime sleep efficiency (i.e., mean percent of time in bed spent asleep) will be calculated from 7 days of wrist actigraphy for patients and caregivers. Range from 0 to 100% with a higher percent indicating better objective sleep quality
Pittsburgh Sleep Quality Index score | immediately after the last session of the intervention
  Self-reported sleep quality over the past week for patients (reported by caregivers) and caregivers. Range from 0 to 21 with lower scores indicating better subjective sleep quality.

SECONDARY OUTCOMES:
Total scores on the Cornell Scale for Depression in Dementia | immediately after the last session of the intervention
  Total scores on the Cornell Scale for Depression in Dementia. Range from 0 to 38 with higher scores indicating worse depressive symptoms among persons with dementia
Total scores on the Patient Health Questionnaire-9 | immediately after the last session of the intervention
  Total scores on the Patient Health Questionnaire-9 for caregivers. Range from from 0 to 27 with higher scores indicating worse depressive symptoms among caregivers
Total scores on the Rating Anxiety in Dementia | immediately after the last session of the intervention
  Total scores on the Rating Anxiety in Dementia for patients. Range from 0 to 54 with higher scores indicating worse anxiety among persons with dementia
Total scores on the Generalized Anxiety Disorder-7 | immediately after the last session of the intervention
  Total scores on the Generalized Anxiety Disorder-7 for caregivers. Range from 0 to 21 with higher scores indicating worse anxiety among caregivers

OTHER OUTCOMES:
Attrition rate | immediately after the posttreatment assessment
  Percent of number of dyads who fail to complete the study both during the intervention and at posttreatment will be measured.
Adherence to homework | immediately after the last session of the intervention
  Percent of days that dyad members complete the homework over the course of the intervention program will be measured.
Interventionist adherence | immediately after the last session of the intervention
  Percent of completion of delivery of each component in sessions will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Yeonsu Song, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided